CLINICAL TRIAL: NCT01152190
Title: A Randomized, Double Blind, Placebo-controlled Study to Evaluate the Effect of Tadalafil Once Daily for 8 Weeks on Prostatic Blood Flow and Perfusion Parameters in Men With Signs and Symptoms of Benign Prostatic Hyperplasia
Brief Title: A Study in Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 13469; H6D-MC-LVIR (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-06-25; First posted 2010-06-29 (Estimated); Results first posted 2013-05-20 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-03

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5 milligrams (mg) Tadalafil (Experimental)
  Interventions: Drug: Tadalafil
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tadalafil — Administered orally, once daily for 8 weeks
  Other Names: Cialis; LY450190
  Arms: 5 milligrams (mg) Tadalafil
Drug: Placebo — Administered orally, once daily for 8 weeks
  Arms: Placebo

SUMMARY:
The purpose of this trial is to evaluate the effect of tadalafil 5 milligrams (mg) daily for 8 weeks compared to placebo on prostatic blood perfusion in men with signs and symptoms of Benign Prostatic Hyperplasia (BPH), measured by resistive index (RI) in the prostate transition zone.

ELIGIBILITY:
Inclusion Criteria

* Present with benign prostatic hyperplasia
* Provide signed informed consent at the screening
* Agree not to use other treatment for Benign Prostatic Hyperplasia, Erectile Dysfunction or Overactive Bladder (including herbal treatments) during the study

Exclusion Criteria

* Have prostatic cancer or are being treated for cancer.
* Any condition that may negatively influence the transrectal ultrasound.
* Are being treated for heart disease with any drug that is called a nitrate (for example, nitroglycerin).
* Any evidence of moderate to severe cardiac disease
* Have had any of the following in the past 90 days: chest pain (called unstable angina or angina) that requires treatment, heart attack also known as myocardial infarction, heart bypass surgery (called coronary artery bypass graft surgery), had a procedure to open up blood vessels in the heart know as angioplasty or stent placement (percutaneous coronary intervention), positive cardiac stress test without effective cardiac intervention.
* Have very high or very low blood pressure.
* Have uncontrolled diabetes.
* Have certain problems with your kidneys, liver, or nervous system.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2010-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Garden City, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Innsbruck, Austria
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bergamo, Italy

REFERENCES:
- [Derived] Pinggera GM, Frauscher F, Paduch DA, Bolyakov A, Efros M, Kaminetsky J, Da Pozzo L, Esler A, Cox D. Effect of tadalafil once daily on prostate blood flow and perfusion in men with lower urinary tract symptoms secondary to benign prostatic hyperplasia: a randomized, double-blind, multicenter, placebo-controlled trial. Urology. 2014 Aug;84(2):412-9. doi: 10.1016/j.urology.2014.02.063. Epub 2014 Jun 14. PMID 24938580

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo: tablet administered orally, once daily for 8 weeks.
- Tadalafil: Tadalafil: 5-milligram (mg) tablet administered orally, once daily for 8 weeks.
Period: Overall Study
Arm/Group | Placebo | Tadalafil
Started | 50 | 47
Received at Least 1 Dose of Study Drug | 50 | 47
Completed | 45 | 39
Not Completed | 5 | 8
Not completed — Adverse Event | 2 | 4
Not completed — Death | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Population: The Primary Analysis Population was defined as all randomized participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tadalafil | Total
Number analyzed (Participants) | 50 | 47 | 97
Age Continuous [Mean (Standard Deviation); unit: years] | 60.3 (8.18) | 60.0 (7.53) | 60.2 (7.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 50 | 47 | 97
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 50 | 45 | 95
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 3 | 11
  White | 41 | 42 | 83
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Austria | 6 | 7 | 13
  Belgium | 4 | 5 | 9
  Italy | 15 | 14 | 29
  United States | 25 | 21 | 46
Erectile Dysfunction (ED) Etiology [Number; unit: participants] — Investigator-reported etiology of a participant's ED at baseline. ED was defined as a consistent change in the quality of an erection adversely affecting the participant's satisfaction with sexual intercourse. ED etiology (psychogenic, organic, mixed, or unknown) was based on the investigator's opinion. Only randomized participants with ED at baseline were summarized (Placebo N=33 and Tadalafil N=29).
  participants
    Psychogenic | 0 | 0 | 0
    Organic | 18 | 15 | 33
    Mixed | 13 | 12 | 25
    Unknown | 2 | 2 | 4
ED Severity [Number; unit: participants] — Investigator-reported severity of a participant's ED at baseline. ED was defined as a consistent change in the quality of an erection adversely affecting the participant's satisfaction with sexual intercourse. The severity (mild, moderate, or severe) of ED was based on the investigator's opinion. Only randomized participants with ED at baseline were summarized (Placebo N=33 and Tadalafil N=29).
  participants
    Mild | 11 | 9 | 20
    Moderate | 16 | 15 | 31
    Severe | 6 | 5 | 11
ED Duration [Number; unit: participants] — Participant-reported ED duration (<1 year or ≥1 year). ED was defined as a consistent change in the quality of an erection adversely affecting the participant's satisfaction with sexual intercourse. Only randomized participants with ED at baseline, who had a baseline ED duration assessment, were summarized (Placebo N=32 and Tadalafil N=29).
  participants
    <1 year | 4 | 1 | 5
    ≥1 year | 28 | 28 | 56
Body Mass Index [Mean (Standard Deviation); unit: kilograms per meter-squared (kg/m^2)] — Body mass index was an estimate of body fat based on body weight divided by height squared.
  kilograms per meter-squared (kg/m^2) | 27.4 (3.19) | 26.4 (3.28) | 26.9 (3.25)
Sitting Diastolic Blood Pressure [Mean (Standard Deviation); unit: millimeters of mercury (mm Hg)] | 81.8 (8.73) | 81.5 (6.85) | 81.7 (7.83)
Sitting Systolic Blood Pressure [Mean (Standard Deviation); unit: millimeters of mercury (mm Hg)] | 131.0 (13.69) | 131.7 (11.96) | 131.4 (12.82)
Baseline Lower Urinary Tract Symptoms (LUTS) Severity [Number; unit: participants] — LUTS was reported as moderate [International Prostate Symptom Score (IPSS) Total Score <20] or severe (IPSS Total Score ≥20). The IPSS Total Score was the sum of Questions 1 through 7 in the IPSS questionnaire. Each question was scored from 0 (none/no symptoms) to 5 (frequent symptoms) for an IPSS Total Score ranging from 0 to 35 points; higher numerical scores from the IPSS questionnaire represented a greater severity of symptoms.
  participants
    Moderate | 22 | 20 | 42
    Severe | 28 | 27 | 55
Urinary Peak Flow Rate (Qmax) [Mean (Standard Deviation); unit: milliliters per second (mL/sec)] — Qmax was measured in mL/sec using a standard, calibrated flowmeter. Only randomized participants with a valid uroflowmetry assessment at baseline were summarized (Placebo N=48 and Tadalafil N=45).
  milliliters per second (mL/sec) | 9.6 (2.50) | 10.4 (2.78) | 10.0 (2.65)
Postvoid Residual Volume [Mean (Standard Deviation); unit: milliliters (mL)] — Postvoid residual volume of urine measured by ultrasound.
  milliliters (mL) | 59.0 (59.11) | 47.8 (44.47) | 53.6 (52.56)
Prostate Specific Antigen [Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)] | 1.9 (1.70) | 2.1 (1.93) | 2.0 (1.81)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 8-Week Endpoint in Arterial Resistive Index (RI) in the Prostate Transition Zone
Description: Arterial RI was a measure of vascular resistance using Doppler ultrasound. RI was the ratio of (peak systolic velocity - end diastolic velocity)/peak systolic velocity, and increased as resistance to blood flow increased. The least squares (LS) mean was estimated from a mixed-effects model with repeated measures (MMRM) that included fixed effects for treatment, region, visit, and treatment-by-visit interaction, baseline as a covariate, a random effect of participant within treatment, and an unstructured covariance matrix.
Time Frame: Baseline, Week 8
Population: Randomized participants who received at least 1 dose of study medication, had non-missing data (arterial RI in the prostate transition zone) at baseline, and a post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 43 | 38
ratio | -0.01 (0.006) | 0.00 (0.006)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.121, Mixed-Model Repeated Measures — The p-value associated with the LS mean difference of change from baseline to Week 8 between the tadalafil and placebo treatment groups was tested at a significance level of 0.05 with no adjustments for multiplicity; Difference in LS Means = 0.01, Standard Error of Mean 0.009

2. Secondary Outcome: Change From Baseline to 4-Week Endpoint in Arterial Resistive Index (RI) in the Prostate Transition Zone
Description: Arterial RI was a measure of vascular resistance using Doppler ultrasound. RI was the ratio of (peak systolic velocity - end diastolic velocity)/peak systolic velocity, and increased as resistance to flow increased. The least squares (LS) mean was estimated from a mixed-effects model with repeated measures (MMRM) that included fixed effects for treatment, region, visit, and treatment-by-visit interaction, baseline as a covariate, a random effect of participant within treatment, and an unstructured covariance matrix.
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 45 | 43
ratio | 0.00 (0.006) | 0.01 (0.006)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.226, Mixed-Model Repeated Measures — The p-value associated with the LS mean difference of change from baseline to Week 4 between the tadalafil and placebo treatment groups was tested at a significance level of 0.05 with no adjustments for multiplicity; Difference in LS Means = 0.01, Standard Error of Mean 0.008

3. Secondary Outcome: Change From Baseline to 4 and 8 Weeks in Arterial Resistive Index (RI) in the Prostate Peripheral Zone and Bladder Neck
Description: as for outcome 2
Time Frame: Baseline, Week 4 and Week 8
Population: Randomized participants who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 45 | 43
ratio
  Week 4 Change, Prostate Peripheral Zone (n=45, 43) | 0.00 (0.006) | 0.01 (0.007)
  Week 8 Change, Prostate Peripheral Zone (n=43, 38) | -0.01 (0.006) | 0.01 (0.007)
  Week 4 Change, Bladder Neck (n=30, 30) | -0.01 (0.012) | 0.01 (0.012)
  Week 8 Change, Bladder Neck (n=32, 26) | 0.01 (0.015) | 0.02 (0.016)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.208, Mixed-Model Repeated Measures — The p-value associated with the LS mean difference of change from baseline to Week 4 in the prostate peripheral zone RI was tested at a significance level of 0.05 with no adjustments for multiplicity; Difference in LS Means = 0.01, Standard Error of Mean 0.009
Statistical Analysis 2: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.066, Mixed-Model Repeated Measures — The p-value associated with the LS mean difference of change from baseline to Week 8 in the prostate peripheral zone RI was tested at a significance level of 0.05 with no adjustments for multiplicity; Difference in LS Means = 0.02, Standard Error of Mean 0.009
Statistical Analysis 3: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.195, Mixed-Model Repeated Measures — The p-value associated with the LS mean difference of change from baseline to Week 4 in bladder neck RI was tested at a significance level of 0.05 with no adjustments for multiplicity; Difference in LS Means = 0.02, Standard Error of Mean 0.017
Statistical Analysis 4: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.625, Mixed-Model Repeated Measures — The p-value associated with the LS mean difference of change from baseline to Week 8 in bladder neck RI was tested at a significance level of 0.05 with no adjustments for multiplicity; Difference in LS Means = 0.01, Standard Error of Mean 0.022

4. Secondary Outcome: Change From Baseline to 4 and 8 Weeks in Color Pixel Intensity (CPI) in the Prostate Transition Zone, Peripheral Zone, and Bladder Neck
Description: CPI quantified blood flow in a pre-specified region of interest by using color Doppler imaging. CPI was the mean color pixel intensity in the region of interest and scores could range from 0 to 160. An increase in CPI reflected an increase in blood flow. The least squares (LS) mean was estimated from a mixed-effects model with repeated measures (MMRM) that included fixed effects for treatment, region, visit, and treatment-by-visit interaction, baseline as a covariate, a random effect of participant within treatment, and an unstructured covariance matrix.
Time Frame: Baseline, Week 4 and Week 8
Population: Randomized participants who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 44 | 43
units on a scale
  Week 4 Change, Prostate Transition Zone (n=44, 43) | -2.21 (2.377) | 0.42 (2.408)
  Week 8 Change, Prostate Transition Zone (n=43, 38) | 2.02 (1.974) | 2.53 (2.083)
  Week 4 Change, Prostate Peripheral Zone (n=44, 43) | -1.48 (2.059) | 1.99 (2.091)
  Week 8 Change, Prostate Peripheral Zone (n=43, 38) | 3.11 (1.868) | 2.55 (1.987)
  Week 4 Change, Bladder Neck (n=42, 40) | 7.37 (4.022) | 3.17 (4.140)
  Week 8 Change, Bladder Neck (n=38, 36) | -0.13 (3.622) | 7.81 (3.738)
Statistical Analysis 1: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.439, Mixed-Model Repeated Measures — The p-value associated with the LS mean difference of change from baseline to Week 4 in the prostate transition zone CPI was tested at a significance level of 0.05 with no adjustments for multiplicity; Difference in LS Means = 2.63, Standard Error of Mean 3.380
Statistical Analysis 2: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.860, Mixed-Model Repeated Measures — The p-value associated with the LS mean difference of change from baseline to Week 8 in the prostate transition zone CPI was tested at a significance level of 0.05 with no adjustments for multiplicity; Difference in LS Means = 0.51, Standard Error of Mean 2.867
Statistical Analysis 3: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.240, Mixed-Model Repeated Measures — The p-value associated with the LS mean difference of change from baseline to Week 4 in the prostate peripheral zone CPI was tested at a significance level of 0.05 with no adjustments for multiplicity; Difference in LS Means = 3.47, Standard Error of Mean 2.937
Statistical Analysis 4: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.839, Mixed-Model Repeated Measures — The p-value associated with the LS mean difference of change from baseline to Week 8 in the prostate peripheral zone CPI was tested at a significance level of 0.05 with no adjustments for multiplicity; Difference in LS Means = -0.55, Standard Error of Mean 2.729
Statistical Analysis 5: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.468, Mixed-Model Repeated Measures — The p-value associated with the LS mean difference of change from baseline to Week 4 in the bladder neck CPI was tested at a significance level of 0.05 with no adjustments for multiplicity; Difference in LS Means = -4.20, Standard Error of Mean 5.770
Statistical Analysis 6: Comparison: Placebo vs Tadalafil; Test type: Superiority or Other; p = 0.131, Mixed-Model Repeated Measures — The p-value associated with the LS mean difference of change from baseline to Week 8 in the bladder neck CPI was tested at a significance level of 0.05 with no adjustments for multiplicity; Difference in LS Means = 7.93, Standard Error of Mean 5.199

ADVERSE EVENTS:
Arm/Group | Placebo | Tadalafil
Serious Adverse Events (participants affected / at risk) | 2/50 | 0/47
Other Adverse Events (participants affected / at risk) | 4/50 | 10/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=50) | Tadalafil (N=47)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) — This event resulted in death.
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=50) | Tadalafil (N=47)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 4 (4)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The primary and secondary efficacy analyses of resistive index (RI) and color pixel intensity (CPI) were based on centrally-read data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days